CLINICAL TRIAL: NCT01547351
Title: Assessing Relapse in Multiple Sclerosis (ARMS) Questionnaire - A Phase 4 Pilot Study
Brief Title: Assessing Relapse in Multiple Sclerosis (ARMS) Questionnaire
Acronym: ARMS
Status: Completed | Type: Observational
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Other Study IDs: QSC02-ARMS-01
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Relapse in multiple sclerosis; Psychometric properties of the patient self-report questionnaire; Evaluation of ARMS questionnaire
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ARMS Questionnaire Group: Patients with confirmed multiple sclerosis relapse who are willing to participate in the ARMS questionnaire. These patients could not have been treated with any therapies other than oral or intravenous corticosteroids for their previous relapse.
  Interventions: Other: ARMS Questionnaire

INTERVENTIONS:
Other: ARMS Questionnaire — The ARMS Questionnaire is a 2-part, 2-page survey, with each part comprising 7 questions on 1 page. Eligible patients will be administered part 1 of the survey when the patient presents with new relapse. Part 2 of the survey is to be completed 1 month (± 1 week) after initiation of treatment for relapse.

SUMMARY:
This Phase 4 pilot cross-sectional descriptive/exploratory study is to be conducted in clinical practice settings (including MS (Multiple sclerosis) specialty clinics, general neurology practices, or other academic or private practice settings) in the United States to assess the psychometric properties of the ARMS questionnaire in approximately 100 adult patients with MS who are experiencing a confirmed relapse, as identified by the investigator or designee at each site. Neither efficacy nor safety of treatment will be evaluated in this study.

The ARMS questionnaire is a 2-part, 2-page survey, with each part comprising 7 questions on 1 page. Part 1 is designed to evaluate the patient's relapse symptoms and how the symptoms affect daily activities and overall function, as well as patient's response to past treatments for previous relapses, as a means of guiding treatment selection. Part 2 is designed to evaluate treatment response in terms of symptom relief and functioning, as well as treatment tolerability. Part 1 of the survey is to be completed when the patient presents with new relapse of MS. Part 2 of the survey is to be completed 1 month (± 1 week) after initiation of treatment for relapse of MS. Treatment for relapse will be at the sole discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and HIPAA authorization must be obtained from the patient prior to any study-related procedures.
* Patient is ≥ 18 years of age at the time of participation
* Patient has confirmed MS relapse.
* Patient must have been treated with oral or IV corticosteroids for their previous relapse.
* Willingness to comply with all procedures and assessments.

Exclusion Criteria:

* Patient has pseudorelapse.
* Patient was treated with any therapies other than corticosteroids for their previous relapse.
* Any other condition which, in the opinion of the investigator, would not allow proper completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practice setting, including academic medical centers and private practices in the US
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total Composite Score (TCS) | After relapse treatment (1 month ± 1 week)
  Total composite score is calculated from three interrelated questions on part 2 of the ARMS questionnaire (to be completed 1 month ± 1 week after relapse treatment).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Tanner Center and Foundation for MS, Birmingham, Alabama
  - Neurology Center, Oceanside, California
  - Infinity Clinical Research, Hollywood, Florida
  - McCare Center Neurology Services, Orlando, Florida
  - Neurology Center of Fairfax, Fairfax, Virginia